CLINICAL TRIAL: NCT07201935
Title: Hot, Cold, and Combined Thermodynamic Exposure to Improve Sleep Quality and Sleep-Time Glymphatic Clearance Among Military Cadets
Brief Title: Thermodynamic Exposure and Sleep in Military Cadets
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00147353
Record Dates: First submitted 2025-09-12; First posted 2025-10-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cold-water Immersion; High Heat Sauna; Combination of Cold-water Immersion and High Heat Sauna
Keywords: Glymphatic System; Sleep quality; Sleep architecture; Thermodynamic exposure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold-water immersion (Experimental): 5 minutes of cold-water immersion (submerged up to chin) at 8 - 10C°(46.4 - 50F°) in the morning between 6:00 - 8:00am.
  Interventions: Behavioral: Cold Water Immersion
- High heat sauna (Experimental): 20 minutes of high heat sauna at 90 - 94C° (190 - 201.2F°) between 5:00 - 7:00pm
  Interventions: Behavioral: High Heat Sauna
- Combination (Experimental): 5 minutes of cold-water immersion (submerged up to chin) at 8 - 10C°(46.4 - 50F°) in the morning between 6:00 - 8:00am and 20 minutes of high heat sauna at 90 - 94C° (190 - 201.2F°) between 5:00 - 7:00pm
  Interventions: Behavioral: Cold Water Immersion; Behavioral: High Heat Sauna

INTERVENTIONS:
Behavioral: Cold Water Immersion — Participants will complete 14 daily sessions of cold-water immersion exposure.
  Arms: Cold-water immersion; Combination
Behavioral: High Heat Sauna — Participants will complete 14 evening sessions in the high heat sauna
  Arms: Combination; High heat sauna

SUMMARY:
This pilot study investigates the effects of cold-water immersion, traditional sauna use, and their combination on sleep architecture, glymphatic clearance, and psycho-affective health in military cadets. The study uses wearable technologies including the Oura Ring and the Applied Cognition Glymphatic Monitor to collect objective sleep and physiological data.

DETAILED DESCRIPTION:
The study will enroll 45 military cadets from The Citadel Military College, randomized into three groups: Cold-Water Immersion (CWI), High Heat Sauna (HHS), and Combined (COM). Participants will undergo a 7-day baseline period followed by a 14-day intervention. Sleep architecture, glymphatic function, and psycho-affective health will be assessed using validated wearable devices and questionnaires. The study aims to identify intervention-specific improvements in sleep and glymphatic clearance.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years of age
* Member of the Ranger Challenge group at The Citadel.
* Access to a smartphone with access to appropriate app marketplace (Apple iOS 15, Android 8.0 or newer) and reliable data access.
* Ability to access and operate Oura Ring application

Exclusion Criteria:

* Medical contraindications to continuous wearing of the Oura Ring.
* Current diagnosis of neurological, cardiovascular, and/or sleep disorder.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Glymphatic clearance | End of baseline monitoring phase (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Changes in parenchymal resistance during sleep
Sleep Efficiency | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Percentage of sleep period spent asleep measured by the Oura Ring (percentage, %)
Pittsburgh Sleep Quality Index | At the end of the baseline monitoring phase (Day 7), end of intervention week 1 (Day 14), and end of intervention phase (Day 28)
  Self-reported sleep quality
Profile of Mood States: Total Mood Disturbance | At the end of the baseline monitoring phase (Day 7), end of intervention week 1 (Day 14), and end of intervention phase (Day 28)
  Self-reported mood disturbance used by summing all negative profiled mood sub-scores (tension, depression, anger/hostility, fatigue, and confusion) and subtracting the positive profiled mood sub-score (vigor). (score -32 - 200, higher equals greater mood disturbance)

SECONDARY OUTCOMES:
Total Sleep Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Total duration of sleep period measured by the Oura Ring (seconds, s)
REM Sleep Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Duration of sleep period spent in REM sleep measured by the Oura Ring (seconds, s)
Deep Sleep Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Duration of sleep periods spent in deep (N3) sleep (seconds, s)
Light Sleep Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Duration of sleep period spent in light (N1 or N2) sleep (seconds, s)
Restless Sleep Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Duration of sleep period with increased registered movements as measured by the Oura Ring (seconds, s)
Wake After Sleep Onset (WASO) Duration | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Total time spent awake after falling asleep (seconds, s)
RMSSD | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Root mean squared of temporal latency between successive heart beats throughout sleep period measured by the Oura Ring (milliseconds, ms)
Nighttime Skin Temperature | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Skin temperature (degrees Celsius, C°) throughout sleep period measured by the Oura Ring.
Profile of Mood States: Tension/Anxiety | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28).
  Tension/Anxiety sub-score computed from the POMS (score 0 - 36, higher equals more tension/anxiety)
Profile of Mood States: Depression | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Depression sub-score from the POMS (score 0 - 60, higher equals greater depression)
Profile of Mood States: Anger/Hostility | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Anger/Hostility sub-score from the POMS (score 0 - 48, higher equals greater anger/hostility)
Profile of Mood States: Vigor | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Vigor sub-score from the POMS (score 0 - 32, higher equals more vigor)
Profile of Mood States: Fatigue | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Fatigue sub-score from the POMS (score 0 - 28, higher equals more fatigue)
Profile of Mood States: Confusion | End of baseline monitoring period (Day 7), end of intervention week 1 (Day 14), and end of intervention (Day 28)
  Confusion sub-score from the POMS (score 0 - 28, higher equals more confusion)
Sleep Time Heart Rate | Each night of the baseline monitoring period (7days) and intervention phase (14days)
  Average heart rate during sleep (beats per minute, bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosenberg, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- The Citadel Military College, Charleston, South Carolina, United States